CLINICAL TRIAL: NCT04582344
Title: Randomized, Double-Blind, Placebo-Controlled Phase III Clinical Trial For Evaluation of Efficacy and Safety of SARS-CoV-2 Vaccine (Vero Cell), Inactivated
Brief Title: Clinical Trial For SARS-CoV-2 Vaccine (COVID-19)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 9026-ASI
Record Dates: First submitted 2020-10-01; First posted 2020-10-09 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2022-08

CONDITIONS: COVID-19
Keywords: COVID-19, SARS-CoV-2 Vaccine
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled Phase III Clinical Trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SARS-COV-2 Vaccine (Experimental): 600 SU of SARS-CoV-2 virus antigen, intramuscular injection, two doses given 14 days apart.
  Interventions: Biological: CoronaVac
- Placebo (Placebo Comparator): Aluminium hydroxide, disodium hydrogen phosphate, sodium dihydrogen phosphate, sodium chloride 0.5mL/dose, intramuscular injection, two doses given 14 days apart.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CoronaVac — Two doses at 14-day interval, each inoculation dose is 0.5 mL. Two doses of dosage (each prefilled syringe of the vaccine contains 600 SU of SARS-CoV-2 virus antigen) experimental vaccine at the schedule of day 0,14
  Arms: SARS-COV-2 Vaccine
Biological: Placebo — Aluminium hydroxide, disodium hydrogen phosphate, sodium dihydrogen phosphate, sodium chloride 0.5mL/dose, two doses given 14 days apart.
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blinded, and placebo controlled phase III clinical trial of the SARS-CoV-2 inactivated vaccine manufactured by Sinovac Research & Development Co., Ltd. The purpose of this study is to evaluate the efficacy, safety and immunogenicity of the experimental vaccine in healthy adults aged 18~59 Years.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded, multi-center, placebo-controlled phase III clinical trial in adults aged 18~59 years. The purpose of this study is to evaluate the efficacy, safety and immunogenicity of the experimental SARS-CoV-2 inactivated vaccine. The experimental vaccine and placebo were both manufactured by Sinovac Research & Development Co., Ltd. A total of 13.000 subjects will be enrolled. Participant will be assigned to receive two doses of experimental vaccine or placebo on the schedule of day 0,14. It is planned that the study will be conducted with two separate cohorts. The first cohort will be healthcare workers in the high risk group (K-1) and the second cohort will be people at normal risk (K-2). After 2 doses of vaccination of 1300 volunteers are completed, safety data will be evaluated by the data safety monitoring board without breaking the blinding, and if there is no safety issue, the K2 cohort will continue to be vaccinated.1.300 volunteers, including 650 volunteers SARS-CoV-2 vaccine and placebo arms, will be included in the K-1 cohort. In the K-2 cohort (normal risk group for COVID-19), 7.650 volunteers were planned to be included in the SARS-CoV-2 vaccine group, and 3.500 volunteers in the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* 18-59 years of age (including 18 and 59 years of ages),
* For only K1 cohort, health care workers such as medical doctor, nurse, ward boy, cleaner, hospital technician, administrative personnel who work in any department of a hospital.
* Signed informed consent

Exclusion Criteria:

* Previously PCR positive for COVID-19
* IgG or IgM is positive
* For females: Pregnancy (confirmed by positive beta-hCG test), breastfeeding or intent to engage in sexual relations with reproductive intent without use of birth control methods in the three months following vaccination
* Known allergy to components of the study vaccine or control
* Use of immunosuppressant therapy regimens within the six months prior to enrollment in the study or planned use within the two years following enrollment. Immunosuppressant therapy regimens include: antineoplastic chemotherapy, radiation therapy and immunosuppressants to induce transplant tolerance, among others
* Use of immunosuppressive doses of corticosteroids within the three months prior to the enrollment in the study and planned use of immunosuppressive doses of corticoids within the three months following enrollment in the study. Immunosuppressive doses of corticosteroids will be considered the equivalent prednisone 20 mg/day for adults, for longer than one week. Continued use of topical or nasal corticosteroids is not considered an immunosuppressant
* History of asplenia
* History of bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture
* Any alcohol or drug abuse over the 12 months prior to enrollment in the study that has caused medical, professional or family problems, indicated by clinical history
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Participation in another clinical trial with an investigational product in the six months prior to enrollment in the study or planned participation in another clinical trial within the two years following enrollment
* Received live attenuated virus vaccine 14 days prior to enrollment in the study
* Inactivated vaccine or sub unit vaccine 7 days prior to enrollment in the study
* Fever (oral temperature >37.2℃, axillary temperature will not be accepted) within the past 24 hours
* Any other condition that, in the opinion of the principal investigator or his/her representative physician, could put the safety/rights of potential participants at risk or prevent them from complying with this protocol.
* Any confirmed or suspected autoimmune disease or immunodeficiency disease, including human immunodeficiency virus (HIV) infection.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10214 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Protection Indexes of Two Vaccine Doses For Symptomatic COVID-19 | 2 weeks after the second dose of vaccination
  The protection rate of a two-dose of SARS-CoV-2 (Vero Cell) vaccine against RT-PCR confirmed symptomatic COVID-19

SECONDARY OUTCOMES:
Protection Indexes of One Vaccine Dose For Symptomatic COVID-19 | 2 weeks after the second dose of vaccination
  The protection rate of, at least, one dose of SARS-CoV-2 (Vero Cell) vaccine against RT-PCR confirmed symptomatic COVID-19 Two weeks after the last dose vaccination.
Protection Indexes of Second Vaccine Dose For Hospitalization, Disease Severity/and Death | 2 weeks after the second dose of vaccination
  The protection rate of a two-dose of SARS-CoV-2 (Vero Cell) vaccine against rates of hospitalization, disease severity/and death two weeks after the second dose of vaccination
Protection Indexes of Two Vaccine Doses For SARS-CoV-2 infection | 2 weeks after the second dose of vaccination
  The protection rate of a two dose of SARS-CoV-2 (Vero Cell) vaccine against RT-PCR confirmed SARS-CoV-2 infection two weeks after the second dose of vaccination
Safety indexes of adverse reactions in 28 days | 28 days after the second dose of vaccination
  The incidence of adverse reactions from the day of first vaccination to 28 days after the second dose of vaccination.
Safety indexes of adverse reactions in 7 days | 7 days after each dose of vaccination
  The incidence of adverse reactions within 7 days after each dose of vaccination
Safety indexes of serious adverse events in 1 year | 1 year after second dose of vaccination
  The incidence of SAEs from the first vaccination to one year after the second dose vaccination
Immunogenicity parameters (seroconversion rate, seropositivity rate) in 14 days | 14 days after each dose vaccination
  The seroconversion rate, seropositivity rate 14 days after each dose vaccination
Immunogenicity parameters (seroconversion rate, seropositivity rate) in 28 days | 28 days after the second dose vaccination
  The seroconversion rate, seropositive rate 28 days after the second dose vaccination
Immunogenicity parameters (GMT and GMI of neutralizing antibody and IgG) in 14 days | 14 days after each dose vaccination
  GMT and GMI of neutralizing antibody and IgG 14 days after each dose vaccination
Immunogenicity parameters (GMT and GMI of neutralizing antibody and IgG) in 28 days | 28 days after the second dose vaccination
  GMT and GMI of neutralizing antibody and IgG 28 days after the second dose vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Murat Akova, Prof., Principal Investigator — Faculty Member
Locations (25):
- Turkey (Türkiye) (25):
  - T.R. Ministry of Health Ankara City Hospital, Infectious Diseases and Clinical Microbiology Clinic, Ankara, Turkey Region
  - T.R. Ministry of Health Ankara Provincial Health Directorate Ankara Training and Research Hospital, Infectious Diseases, Ankara, Turkey Region
  - Ankara University Faculty of Medicine, Department of Infectious Diseases and Clinical Microbiology, Ankara, Turkey Region
  - Çukurova University Faculty of Medicine, Department of Infectious Diseases, Adana
  - Hacettepe University Faculty of Medicine Department of Infections Diseases and Clinical Microbiology, Ankara
  - T.C Ministry of Health Ankara Provincial Health Directorate Health Sciences University Ankara Atatürk Chest Diseases and Thoracic Surgery Training and Research Hospital, Ankara
  - Akdeniz University Faculty of Medicine, Department of Infectious Diseases, Antalya
  - Bursa Uludağ University Faculty of Medicine, Department of Infectious Diseases and Clinical Microbiology, Bursa
  - Dicle University Faculty of Medicine, Department of Infectious Diseases and Clinical Microbiology, Diyarbakır
  - Gaziantep University Faculty of Medicine, Department of Infectious Diseases and Clinical Microbiology, Gaziantep
  - Acıbadem Atakent Hospital, Infectious Diseases and Clinical Microbiology, Istanbul
  - Cerrahpaşa Faculty of Medicine, Department of Internal Medicine - Department of Infectious Diseases and Clinical Microbiology, Istanbul
  - Istanbul Medipol University Faculty of Medicine, Department of Internal Medicine, Istanbul
  - Istanbul University Istanbul Faculty of Medicine, Department of Infectious Diseases and Clinical Microbiology, Istanbul
  - T.R. Ministry of Health Istanbul Provincial Health Directorate Marmara Univesity Istanbul Pendik Education and Research Hospital, Istanbul
  - T.R. Ministry of Health Istanbul Provincial Health Directorate Prof. Dr. Cemil Taşçıoğlu City Hospital, Infectious Diseases Clinic, Istanbul
  - T.R. Ministry of Health Istanbul Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital, Istanbul
  - University of Health Sciences İstanbul Ümraniye Training and Research Hospital, Istanbul
  - Ege University Faculty of Medicine Hospital, Department of Infectious Diseasesaculty of Medicine Hospital, Department of Infectious Diseases, Izmir
  - Republic Of Turkey Ministry Of Health Izmir Provincial Health Directorate Health Sciences University Dr Suat Seren Chest Diseases And Chest Surgery Training And Research Hospital, Izmir
  - T.R. Ministry of Health İzmir Provincial Health Directorate İzmir Health Sciences University Tepecik Training and Research Hospital, Infectious Diseases, Izmir
  - T.R. Ministry of Health Kayseri City Training and Research Hospital, Infectious Diseases and Clinical Microbiology Department, Kayseri
  - Kocaeli University Faculty of Medicine, Department of Infectious Diseases and Clinical Microbiology, Kocaeli
  - Malatya İnönü University Faculty of Medicine, Department of Infectious Diseases, Malatya
  - Karadeniz Technical University Medical Faculty Hospital, Department of Infectious Diseases and Clinical Microbiology, Trabzon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gao Q, Bao L, Mao H, Wang L, Xu K, Yang M, Li Y, Zhu L, Wang N, Lv Z, Gao H, Ge X, Kan B, Hu Y, Liu J, Cai F, Jiang D, Yin Y, Qin C, Li J, Gong X, Lou X, Shi W, Wu D, Zhang H, Zhu L, Deng W, Li Y, Lu J, Li C, Wang X, Yin W, Zhang Y, Qin C. Development of an inactivated vaccine candidate for SARS-CoV-2. Science. 2020 Jul 3;369(6499):77-81. doi: 10.1126/science.abc1932. Epub 2020 May 6. PMID 32376603
- [Derived] Luan N, Li T, Wang Y, Cao H, Yin X, Lin K, Liu C. Th2-Oriented Immune Serum After SARS-CoV-2 Vaccination Does Not Enhance Infection In Vitro. Front Immunol. 2022 Apr 8;13:882856. doi: 10.3389/fimmu.2022.882856. eCollection 2022. PMID 35464483
- [Derived] Tanriover MD, Doganay HL, Akova M, Guner HR, Azap A, Akhan S, Kose S, Erdinc FS, Akalin EH, Tabak OF, Pullukcu H, Batum O, Simsek Yavuz S, Turhan O, Yildirmak MT, Koksal I, Tasova Y, Korten V, Yilmaz G, Celen MK, Altin S, Celik I, Bayindir Y, Karaoglan I, Yilmaz A, Ozkul A, Gur H, Unal S; CoronaVac Study Group. Efficacy and safety of an inactivated whole-virion SARS-CoV-2 vaccine (CoronaVac): interim results of a double-blind, randomised, placebo-controlled, phase 3 trial in Turkey. Lancet. 2021 Jul 17;398(10296):213-222. doi: 10.1016/S0140-6736(21)01429-X. Epub 2021 Jul 8. PMID 34246358
- [Derived] Akova M, Unal S. A randomized, double-blind, placebo-controlled phase III clinical trial to evaluate the efficacy and safety of SARS-CoV-2 vaccine (inactivated, Vero cell): a structured summary of a study protocol for a randomised controlled trial. Trials. 2021 Apr 13;22(1):276. doi: 10.1186/s13063-021-05180-1. PMID 33849629